CLINICAL TRIAL: NCT01777828
Title: Registry of Aortic Valve Bioprostheses Established by Catheter
Acronym: FRANCE-TAVI
Status: Recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 12650
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Transcatheter Aortic Valve Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transcatheter Aortic Valve Implantation: FRANCE TAVI registry aims to identify all patients with a change of valves implanted catheter meets the selection criteria of the technical accepting the scheduled evaluations in the context of this disease and who have agreed to participate in the study .

SUMMARY:
The aim of this registry is to evaluate the overall survival up to 10 years of patients with aortic valve bioprostheses implanted via the transarterial or transapical route. Data from the register is enhanced by matching it with continuous data in the SNDS.

Mandated by the French health authorities, this registry must be maintained as part of the management of any patient undergoing transarterial or transapical aortic valve bioprosthesis implantation.

Participation in the registry is offered to all subjects eligible for bioprosthesis implantation.

DETAILED DESCRIPTION:
Aortic valve stenosis is a serious chronic life-threatening in the short or medium term since the onset of functional symptoms. Aortic valve replacement surgery is currently the treatment of choice. It is done by surgery with sternotomy and extracorporeal circulation. However, despite the considerable improvement of the conditions of care per and post operative, this procedure is sometimes burdened with high mortality, especially in the population with severe co-morbidities and / or many. For this reason, some patients are considered against the indicated surgery or high surgical risk.

The recent development of aortic valve bioprostheses implanted with new approaches (pressure or transapical) can be considered for aortic valve replacement in a population that was previously excluded.

Based on very thorough evaluation of these valves test benches and animal as well as human settlements achieved through multiple studies and registries mono or multi patients challenged by cardiac surgeons or considered at high surgical risk, it is clear that the implementation of these valves could allow, under conditions of optimal implementation and monitoring, improve short-and long-term clinical status, quality of life and prognosis of patients.

FRANCE 2 registry, established in 2010, and whose inclusions ended 30 June 2012 has allowed an initial assessment of aortic valve bioprostheses implanted catheter The following registry France 2 has been requested by the highest authorities of health, FRANCE register TAVI is performed in continuity FRANCE 2. It takes account of the first data FRANCE 2. Data Report Form has been reduced, no new item has been added, it will be carried out in all centers authorized in France to implement this technique. The collection of data will TAVI France under the same conditions as those FRANCE 2, the database will be managed by the French Society of Cardiology

ELIGIBILITY:
Inclusion Criteria: Patients who have undergone transarterial or transapical aortic valve bioprosthesis implantation

Exclusion Criteria: Patient has not given consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participation in the registry will be offered to all subjects eligible for bioprosthesis implantation.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2033-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
10 year survival | 10 year
  After leaving the hospital, the doctor responsible for the register in each center will contact annually the patient or his family and referring physicians by phone to take new or fix an appointment for consultation. This data is supplemented by automatic collection through the SNDS link. The study is purely observational, it does not require special monitoring visits but involves collecting data obtained during routine follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes - Pontchaillou, Rennes, France

REFERENCES:
- [Background] Gilard M, Eltchaninoff H, Iung B, Donzeau-Gouge P, Chevreul K, Fajadet J, Leprince P, Leguerrier A, Lievre M, Prat A, Teiger E, Lefevre T, Himbert D, Tchetche D, Carrie D, Albat B, Cribier A, Rioufol G, Sudre A, Blanchard D, Collet F, Dos Santos P, Meneveau N, Tirouvanziam A, Caussin C, Guyon P, Boschat J, Le Breton H, Collart F, Houel R, Delpine S, Souteyrand G, Favereau X, Ohlmann P, Doisy V, Grollier G, Gommeaux A, Claudel JP, Bourlon F, Bertrand B, Van Belle E, Laskar M; FRANCE 2 Investigators. Registry of transcatheter aortic-valve implantation in high-risk patients. N Engl J Med. 2012 May 3;366(18):1705-15. doi: 10.1056/NEJMoa1114705. PMID 22551129
- [Result] Auffret V, Lefevre T, Van Belle E, Eltchaninoff H, Iung B, Koning R, Motreff P, Leprince P, Verhoye JP, Manigold T, Souteyrand G, Boulmier D, Joly P, Pinaud F, Himbert D, Collet JP, Rioufol G, Ghostine S, Bar O, Dibie A, Champagnac D, Leroux L, Collet F, Teiger E, Darremont O, Folliguet T, Leclercq F, Lhermusier T, Olhmann P, Huret B, Lorgis L, Drogoul L, Bertrand B, Spaulding C, Quilliet L, Cuisset T, Delomez M, Beygui F, Claudel JP, Hepp A, Jegou A, Gommeaux A, Mirode A, Christiaens L, Christophe C, Cassat C, Metz D, Mangin L, Isaaz K, Jacquemin L, Guyon P, Pouillot C, Makowski S, Bataille V, Rodes-Cabau J, Gilard M, Le Breton H; FRANCE TAVI Investigators. Temporal Trends in Transcatheter Aortic Valve Replacement in France: FRANCE 2 to FRANCE TAVI. J Am Coll Cardiol. 2017 Jul 4;70(1):42-55. doi: 10.1016/j.jacc.2017.04.053. PMID 28662806
- [Result] Auffret V, Bedossa M, Boulmier D, Verhoye JP, Ruggieri VG, Koning R, Laskar M, Van Belle E, Leprince P, Collet JP, Iung B, Lefevre T, Eltchaninoff H, Gilard M, Le Breton H. [From FRANCE 2 to FRANCE TAVI: are indications, technique and results of transcatheter aortic valve replacement the same?]. Presse Med. 2015 Jul-Aug;44(7-8):752-60. doi: 10.1016/j.lpm.2015.05.004. Epub 2015 Jul 22. French. PMID 26208911
- [Result] Folliguet TA, Teiger E, Beurtheret S, Modine T, Lefevre T, Van Belle E, Gilard M, Eltchaninoff H, Koning R, Iung B, Verhoye JP, Leprince P, Le Breton H, Lafont A, Parolari A, Barili F. Carotid versus femoral access for transcatheter aortic valve implantation: a propensity score inverse probability weighting study. Eur J Cardiothorac Surg. 2019 Dec 1;56(6):1140-1146. doi: 10.1093/ejcts/ezz216. PMID 31365061
- [Result] Benamer H, Auffret V, Cayla G, Chevalier B, Dupouy P, Eltchaninoff H, Gilard M, Guerin P, Iung B, Koning R, Monsegu J, Lantelme P, Le Breton H, Lefevre T, Verhoye JP, Commeau P, Motreff P. Position paper of French Interventional Group (GACI) for TAVI in France in 2018. Ann Cardiol Angeiol (Paris). 2018 Dec;67(6):455-465. doi: 10.1016/j.ancard.2018.09.021. Epub 2018 Oct 28. PMID 30376969
- [Result] Deharo P, Jaussaud N, Grisoli D, Camus O, Resseguier N, Le Breton H, Auffret V, Verhoye JP, Koning R, Lefevre T, Van Belle E, Eltchaninoff H, Gilard M, Leprince P, Iung B, Lambert M, Collart F, Cuisset T. Impact of Direct Transcatheter Aortic Valve Replacement Without Balloon Aortic Valvuloplasty on Procedural and Clinical Outcomes: Insights From the FRANCE TAVI Registry. JACC Cardiovasc Interv. 2018 Oct 8;11(19):1956-1965. doi: 10.1016/j.jcin.2018.06.023. Epub 2018 Sep 12. PMID 30219324
- [Result] Didier R, Gouysse M, Eltchaninoff H, Le Breton H, Commeau P, Cayla G, Glatt N, Glatt B, Gabbas M, Tuppin P, Liepchitz L, Boussac M, Iung B, Gilard M. Successful linkage of French large-scale national registry populations to national reimbursement data: Improved data completeness and minimized loss to follow-up. Arch Cardiovasc Dis. 2020 Aug-Sep;113(8-9):534-541. doi: 10.1016/j.acvd.2020.04.006. Epub 2020 Jul 22. PMID 32712203
- [Derived] Van Belle E, Vincent F, Labreuche J, Auffret V, Debry N, Lefevre T, Eltchaninoff H, Manigold T, Gilard M, Verhoye JP, Himbert D, Koning R, Collet JP, Leprince P, Teiger E, Duhamel A, Cosenza A, Schurtz G, Porouchani S, Lattuca B, Robin E, Coisne A, Modine T, Richardson M, Joly P, Rioufol G, Ghostine S, Bar O, Amabile N, Champagnac D, Ohlmann P, Meneveau N, Lhermusier T, Leroux L, Leclercq F, Gandet T, Pinaud F, Cuisset T, Motreff P, Souteyrand G, Iung B, Folliguet T, Commeau P, Cayla G, Bayet G, Darremont O, Spaulding C, Le Breton H, Delhaye C. Balloon-Expandable Versus Self-Expanding Transcatheter Aortic Valve Replacement: A Propensity-Matched Comparison From the FRANCE-TAVI Registry. Circulation. 2020 Jan 28;141(4):243-259. doi: 10.1161/CIRCULATIONAHA.119.043785. Epub 2019 Nov 16. PMID 31736356